CLINICAL TRIAL: NCT02896959
Title: How Much is Too Much: Assessing Varying Pressure Pump Pressures in Post Operative Pain Control in Shoulder Arthroscopy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 106756
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Shoulder Arthroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 25mmHg pressure (Experimental): Pump pressure of 25mmHg during rotator cuff repair
  Interventions: Procedure: Arthroscopic rotator cuff repair
- 45mmHg pressure (Experimental): Pump pressure of 45mmHg during rotator cuff repair
  Interventions: Procedure: Arthroscopic rotator cuff repair
- 65mmHg pressure (Experimental): Pump pressure of 65mmHg during rotator cuff repair
  Interventions: Procedure: Arthroscopic rotator cuff repair

INTERVENTIONS:
Procedure: Arthroscopic rotator cuff repair

SUMMARY:
Postoperative surgical pain has been extensively study with regard to anaesthesia pain modalities, however little is published with regards to various arthroscopic shoulder surgical techniques. An intriguing characteristic of shoulder arthroscopy is the various arthroscopic pump pressures used by different surgeons. One could hypothesize that excessive water retention from the arthroscopic pump could causes excessive tissue pressure and swelling resulting in post operative pain. Unfortunately we could not find any literature in the English language regarding varying pressure pump settings on post operative pain control. For that reason we would like to assess how variable pump pressure effect tissue pressure over pre set time points, and how this may relate to post operative pain control.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending St. Joseph's hospital
* Shoulder pathology amenable to arthroscopic surgery
* Medically suitable for surgical management
* Able to consent for surgery.

Exclusion Criteria:

* Unable to consent
* Active infection
* Active malignancy
* Drug or alcohol misuse
* Work related injury
* Lack of permanent home residence
* Previous surgery to affected shoulder
* Medical contraindiction to surgery
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Pain - VAS scale | Two years